CLINICAL TRIAL: NCT06269575
Title: Evaluation Of The Effectiveness Of Safe Nutrition Program Applied To Acute Stroke Patients With Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Zeliha Tülek, Prof., Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Dysphagia
Record Dates: First submitted 2024-01-04; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: DYSPHAGIA
Keywords: DYSPHAGIA; STROKE
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Intervention Model Description: non-randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): safe nutrition arm
  Interventions: Behavioral: SAFE NUTRITION PROGRAM
- control arm (No Intervention): control arm

INTERVENTIONS:
Behavioral: SAFE NUTRITION PROGRAM — Safe nutrition program:
  patient education, caregiver training, behavioral swallowing intervention, position, oral care, swallowing exercises, swallowing assessment
  Arms: experimental

SUMMARY:
It was planned in a quasi-experimental design with a non-randomized control group. The study was planned to be completed in three stages: control, preparation and intervention periods.

Question 1: Does a safe nutrition program prevent aspiration pneumonia, dehydration and malnutrition in acute stroke patients with dysphagia? Question 2: Is the safe nutrition program effective on addiction level, quality of life and depression in acute stroke patients with dysphagia? Question 3: Does a safe nutrition program shorten the hospital stay and NG tube duration in acute stroke patients with dysphagia?

DETAILED DESCRIPTION:
Introduction: Dysphagia is a common complication in acute stroke patients. Although there are treatment options, healing takes time. Managing this process in the safest way is important for the physical and mental health of the patient.

Purpose: This study aimed to evaluate the effectiveness of a safe nutrition program applied to acute stroke patients with dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* acute stroke patients
* 18 years and over

Exclusion Criteria:

* those who do not want to be involved in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Complications of dysphagia | 3 months
  aspiration pneumonia
Complications of dysphagia | 3 months
  Dehydration
Complications of dysphagia | 3 months
  malnutrition

SECONDARY OUTCOMES:
Stroke-Specific Quality of Life Scale (SS-QOL) | 3 months
  A high score on the scale indicates a high quality of life, A low score indicates a low quality of life. (Max:235; min: 48)
Swallowing Anxiety Scale (YKÖ) | 3 months
  Getting a high score from the scale indicates that the individual's swallowing anxiety symptoms increase. (max: 40; min: 0)

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Cavusoglu, Principal Investigator — Istanbul Universitesi-Cerrahpasa; Zeliha Tulek, Study Director — Istanbul Universitesi-Cerrahpasa
Locations (1):
- Istanbul Universitesi-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No